CLINICAL TRIAL: NCT03848520
Title: Do People Run Following a TKA? A Cross-sectional Survey Study Addressed to Patients.
Brief Title: Survey of Running Following a TKA
Status: Completed | Type: Observational
Sponsor: Brigitte Jolles, MD (Other)
Responsible Party: Sponsor-Investigator, Brigitte Jolles, MD, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Other Study IDs: 2018-00386
Record Dates: First submitted 2018-06-11; First posted 2019-02-20 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Arthroplasty; Knee Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total Knee Arthroplasty: Internal Registry of Patients having a TKA and with a high (>=9) activity-scale score at anytime between preoperatively and now.
  Interventions: Procedure: TKA

INTERVENTIONS:
Procedure: TKA — TKA performed in the past

SUMMARY:
The hypothesis of this study is that there are people running following a total knee arthroplasty (TKA).

The objective is (1) to determine if there are people that ran/run following their TKA and (2), in case (1) is true, to identify some general running parameters such as duration, frequency, perceived barriers for running.

Patients with a TKA and a score equal or higher than 9 on the UCLA activity scale at any time between 2 years prior to surgery and at present will be invited to participate in the trial by phone. All these patients will receive the study's information form and questionnaire by post with a pre-stamped envelope to return the documents.The survey was created and piloted internally for this study. There are 21 questions, most of them are "yes or no" and some others open questions to assess parameters such as duration of difficulties faced. The questionnaire is composed of three parts. The first part is interested in the preoperative activity (during the 2 years before surgery), the second part in the postoperative activity (during the 2 years after surgery) and the third part refers to the current practice. For each part, people are asked about specific practice parameters and modalities. Furthermore, we seek to determine whether there was/is a willingness to run following TKA, if patients receive any education/information about it and their personal attitudes towards running with a TKA. The anonymized data will be collected by the main author for subsequent analysis.

ELIGIBILITY:
Inclusion Criteria:

* TKA and UCLA score = or > 9

Exclusion Criteria:

* Inability to read/write in french language
* Cognitive or neurological impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Human adults that underwent a TKA at the investigator's Hospital and with data available on the Institution's Implants Registry
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Changes in number of runners following a TKA | From preoperatively to up to 20 years following TKA. From date of the preoperative assessment until the last clinical assessment available following TKA
  Due to the limited number of patients availabe the analysis will be performed through a qualitative questionnaire. It has 21 questions, most of them are "yes or no" choice and some other open to assess parameters such as "number of runners", "frequency of running" (x/week), "duration of running" (min) and "patients' attitudes towards running" (adjectives reported) with a TKA. It is a patient based questionnaire to be send to each patient and returned by post.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No